CLINICAL TRIAL: NCT02284295
Title: Molecular, Cytological Features and Genetic Susceptibility of Occupational Chronic Obstructive Pulmonary Disease Attributable to Different Environmental Exposures 2.
Brief Title: Molecular, Cytological Features and Genetic Susceptibility of COPD Attributable to Different Environmental Exposures 2
Status: Completed | Type: Observational
Sponsor: Novosibirsk City Hospital #2 (Other)
Collaborators: Siberian Branch of the Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Liubov A Shpagina, Prof., Dr, Novosibirsk City Hospital #2
Other Study IDs: 01201463369/2; 01201463369 (Other: Education and Science Ministry of Russian Federation)
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; silica dust; aromatic hydrocarbons; genetic; occupational
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum,bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- occupational COPD: Consists of 2 subgroups
  1. COPD patients with history of exposure to respirable silica dust
  2. COPD patients with history of exposure to aromatic hydrocarbons
  Interventions: Other: exposure to respirable silica dust; Other: exposure to aromatic hydrocarbons
- smokers with COPD and healthy control: 1. patients with COPD, history of tobacco smoke and no history of occupational exposure
  2. healthy subjects

INTERVENTIONS:
Other: exposure to respirable silica dust — History of exposure to respirable silica dust due to job
  Groups: occupational COPD
Other: exposure to aromatic hydrocarbons — history of exposure to aromatic hydrocarbons due to job
  Groups: occupational COPD

SUMMARY:
The objective of this study is to investigate molecular, cytological and genetic features of occupational chronic obstructive pulmonary disease (COPD) in conditions of different occupational exposures. In order to achieve this goal serum pro-inflammatory cytokines and standard inflammation markers level, hemostasis, cytological analysis of bronchoalveolar lavage fluid and association of single nucleotide polymorphisms (SNPs) rs1800470 transforming growing factor β1 (TGF β1) gene, rs1828591 hedgehog interacting protein (HHIP) gene, rs4129267 interleukin 6 receptor (IL-6R) gene, rs1051730 nicotinic acetylcholine receptor 3 (CHRNA3) gene with COPD in subjects exposed to silica dust and in those exposed to polycyclic aromatic hydrocarbons exhaust will be investigated. The relationship between genotype and phenotype characteristics, such as an inflammation activity, assessed by C-reactive protein (hsCRP) and tumor necrosis factor alpha (TNF α) serum concentration, in different occupational COPD groups will be studied. The hypothesis is that the mechanisms underlying disease development and progression are different due to environmental risk factor that reflex in differs in disease attributes - molecular biomarkers, cytology results and genetic susceptibility between COPD due to dust, COPD due to chemicals and COPD in smokers therefore COPD can be subdivided into ecological phenotypes according to environmental risk factor.

DETAILED DESCRIPTION:
Study rationale: The main risk factors of COPD are tobacco smoking, biomass smoking and occupational factors. Tobacco smoking is well-known risk factor so tobacco induced COPD is completely established. Nevertheless the meaning of occupational factors which are less famous are equally important. Based on comprehensive literature review ATS endorsed the notion that strong evidence implicates occupational factors as cause of COPD. Occupational COPD takes 19.2 % of all COPD patients and 31.1 % of never smokers as resulted NHANESIII study. A considerable number of work-related factors have evidence for a causal association with COPD including (and of course not limited) silica and silicates and aromatic hydrocarbons. Individuals in a variety of occupations and industries such as coal miners, painters, coke workers, tunnel workers, metallurgists, welding workers, transportation workers, builders, farmers are exposed to factors cited above. Despite this the clinical and pathophysiological features of COPD caused by occupational factors are still unclear.

Occupational factors leading airflow limitation are various entities - vapors, dusts, gases and fumes with different physical, chemical, biological and other features, so the mechanisms underlying disease development and progression may be different attributable to risk factor.

An environmental risk factors exposure as well as tobacco smoking results in COPD only in part of the subjects which indicates the significant genome and gene environmental interactions role. COPD develops in predisposed subjects undergoing risk factors exposure. Therefore the risk of COPD is individual and depends on both genetic and environments. There are few data concerning the effects of genetic on COPD risk in this specific subgroup - people who are exposed to occupational risk factors related to the certain environmental factor.

Statistical analysis: Statistical analysis will be carried out by Statistica 9.0 software. Significance level will be considered p = 0.05. The qualitative variables will be expressed as counts and percentages. The quantitative continuous variables will be expressed as means and standard error of means (M ± m) for variables that meet the criteria of normality and minimum and maximum, median for those that do not meet the criteria of normality. Kruskal-Wallis test will be used for comparing multiply independent samples and Mann-Whitney U test for comparing two independent samples if variable under consideration will continuous and that it will be measured on an ordinal scale. For comparisons of proportions, the Chi-square will be used.

For associations assessment we will use logistic regression method. The odds ratios (OR) and 95% confidence intervals (CI) will be calculated for each professional group. Multiple regression model will be used to explore the relationships between demographic characteristics, cytokine concentrations, hemostasis and airflow limitation in professional groups.

ELIGIBILITY:
Inclusion Criteria:

* Post- bronchodilator forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) ratio less than 0.7
* Stable phase of COPD
* History of exposure to respirable silica dust, nonsmokers with no of passive exposure of tobacco smoke or history of exposure to aromatic hydrocarbons, nonsmokers with no of passive exposure of tobacco smoke or current tobacco smokers without history of occupational exposure
* COPD risk factor exposure (occupational or tobacco smoke) duration not less than 12 months
* Male
* Caucasian
* Age of 40 - 75 years old

Exclusion Criteria:

* history of biomass smoke exposure
* age less than 40 and above 75 years old
* current COPD exacerbation
* concomitant asthma
* tuberculosis and other pulmonary diseases
* allergic and autoimmune disorders
* active infections
* immunodeficiency, including HIV infection
* parasitological diseases
* malignancies
* lack of informed consent.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of a certain town (Novosibirsk, Russian Federation)
Sampling Method: Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Difference in serum interleukin 1 beta (IL-1β) level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in serum tumor necrosis factor alpha (TNFα) level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in spontaneous thrombocyte aggregation between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in collagen induced thrombocyte aggregation between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in epinephrine induced thrombocyte aggregation between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in adenosine diphosphate induced thrombocyte aggregation between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in fibrinogen level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in fibrinogen degradation products level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in D-dimer level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in serum endothelin1 level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Difference in serum nitric oxide level between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Differences in cytological analysis of bronchoalveolar lavage fluid results between COPD patients exposed to dust, chemicals and tobacco smoke | 1 day (a single measurement)
  Comparison of groups
Association of SNPs rs1800470 TGF β1 gene, rs1828591 HHIP gene, rs4129267 IL-6R gene, rs1051730 CHRNA3 gene with COPD in subjects exposed to dust and in those exposed to chemicals. (Odds ratio and 95% confidence interval) | 1 day (a single measurement)
  Odds ratio and 95% confidence interval will be calculated for each occupational group. Controls - healthy people.

SECONDARY OUTCOMES:
Relationship between genotype and phenotype characteristics, such as an inflammation activity, assessed by hsCRP and TNF α serum concentration, in different occupational COPD groups. | 1 day (a single measurement)
  For SNPs that will occur associated with occupational COPD differences in hsCRP and TNFα serum concentration between subjects with different genotypes will be established separately for exposed to dust COPD group and for exposed to chemicals COPD group.

CONTACTS AND LOCATIONS:
Overall Officials: Liubov Shpagina, PhD, Principal Investigator — Novosibirsk City Hospital #2, Novosibirsk State Medical University
Locations (1):
- Novosibirsk City Hospital #2, Novosibirsk, Russia